CLINICAL TRIAL: NCT02559388
Title: Assessment of Montelukast Efficacy in the Treatment of Refractive Uremic Pruritus
Brief Title: Montelukast for Treatment of Uremic Pruritus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Mahmudpour, Fellowship of Nephrology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SUMS.REC.1394.32
Record Dates: First submitted 2015-09-09; First posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- montelukast (Active Comparator): montelukast 10 milligram, daily for 30 days
  Interventions: Drug: Montelukast
- placebo (Placebo Comparator): Placebo one tablet for 30 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Montelukast
  Arms: montelukast
Drug: placebo — Placebo (For Montelukast) Placebo pills manufactured for mimic 10 milligram montelukast pills
  Arms: placebo

SUMMARY:
In this study hemodialysis patients that underwent dialysis thrice weekly screen for uremic pruritus and 80 patients that at least have refractive pruritus that lead to sleep and daily activity disorders enroll in this study. These patients should have at least a course of therapy without proper response. After proper informing patients and taking testimonial patients enter to study. Then patients randomized in case and control group. In case group, patients took montelukast 10 milligram daily and in control group took placebo for 30 days. Other antipruritic or antiinflammatory medication has been stopped one week prior to starting treatment. Calcium, phosphorous, urea, creatinine, highly sensitive CRP (hsCRP), Parathyroid Hormone (PTH), hemoglobin and kt/V were measured at beginning and at end of study. pruritus severity assessed by Detailed Pruritus Score that introduced by Duo and Visual Analogue Score in beginning and at end of study in both group. Sleep disorder score and its severity added to crude score at beginning and end of study and change of measures analyzed.

DETAILED DESCRIPTION:
Montelukast is an antileukotrien receptor antagonist that seems to be effective as an antipruritic medication via blocking inflammatory pathways.

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis patients that refered to dialysis centers and at least on hemodialysis thrice weekly
* presence of uremic pruritus
* patients that at least had refractive pruritus that lead to sleep disorders or compromised daily activities
* patients should took a course of antipruritic treatment with no proper response

Exclusion Criteria:

* presence of pruritus less than three months
* kt/V less than 1.2
* presence of pruritus due to other cause other than uremic state
* presence of other pruritic diseases; malignancies; cholestasis; hepatitis B and C infection
* treatment with corticosteroid
* presence of anemia with hemoglobin less than 10

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Detailed score proposed by Duo for pruritus | Change from Baseline in Detailed score at 1months
  Change from Baseline in Detailed score at 1months

SECONDARY OUTCOMES:
Highly sensitive CRP (hs-CRP) | Change from Baseline in serum value at 1months
  This test is a serologic biochemical test

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Mehdi Sagheb, Professor, Principal Investigator — Shiraz University of Medical Sciences

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264